CLINICAL TRIAL: NCT02835118
Title: A Randomized, Double-Blinded, Placebo-Controlled, Multiple-Dose, Safety and Pharmacokinetic Study of Ascending Doses of Oral CB-183,315 in Healthy Volunteers
Brief Title: A Study of Ascending Multiple Doses of Oral Surotomycin in Healthy Participants (MK-4261-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4261-009
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Clostridium Difficile Associated Diarrhea (CDAD)
MeSH Terms: interventions — CB-183,315

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Surotomycin 0.5 g (Experimental): Two oral doses of 0.25 g surotomycin in hard gelatin capsules per day, taken at least 8 hours apart, for 14 days
  Interventions: Drug: Surotomycin
- Surotomycin 1 g (Experimental): Two oral doses of 0.5 g surotomycin in hard gelatin capsules per day, taken at least 8 hours apart, for 14 days
  Interventions: Drug: Surotomycin
- Surotomycin 2 g (Experimental): Two oral doses of 1 g surotomycin in hard gelatin capsules per day, taken at least 8 hours apart, for 14 days
  Interventions: Drug: Surotomycin
- Placebo (Placebo Comparator): Two oral doses of placebo for surotomycin in hard gelatin capsules per day, taken at least 8 hours apart, for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Surotomycin — Two oral doses of surotomycin in hard gelatin capsules totaling either 0.5, 1 or 2 g per day, for 14 days
  Other Names: CB-183,315
  Arms: Surotomycin 0.5 g; Surotomycin 1 g; Surotomycin 2 g
Drug: Placebo — Two oral doses of placebo for surotomycin in hard gelatin capsules per day, for 14 days
  Arms: Placebo

SUMMARY:
This study aims to assess the safety, tolerability, and pharmacokinetics (PK) of oral doses of surotomycin (CB-183,315) administered for 14 consecutive days in healthy males and females.

ELIGIBILITY:
Inclusion Criteria:

* Has no evidence of prior chronic gastrointestinal inflammatory disease such as inflammatory bowel disease
* Electrocardiogram (ECG) shows no clinically significant abnormalities
* Is in good health

Exclusion Criteria:

* Pregnant or lactating females
* Has prior exposure to surotomycin
* Has received an investigational drug or participated in any experimental procedure within1 month prior to study entry and at least 6 half lives from last intake of study drug
* Participants 18 to 49 years of age that has taken any regular, prescribed, or over-the-counter medication
* Has any significant concurrent therapies
* Has a positive drug screen
* Has a positive human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C screen
* Has donated blood or blood products in the 60 days preceding screening
* Is an active intravenous drug user or abuses alcohol
* Has had a malignancy within the last 5 years
* Has inadequate protection against pregnancy during the conduct of the study and until 1 month after last dose of study drug
* Has received any antibiotics within 30 days prior to first dose of study drug
* Has known hypersensitivity to daptomycin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with an Adverse Event (AE) | Up to Day 21
Number of participants who discontinued study treatment due to an AE | Up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Chandorkar G, Zhan Q, Donovan J, Rege S, Patino H. Pharmacokinetics of surotomycin from phase 1 single and multiple ascending dose studies in healthy volunteers. BMC Pharmacol Toxicol. 2017 Mar 28;18(1):24. doi: 10.1186/s40360-017-0123-z. PMID 28347318